CLINICAL TRIAL: NCT01283945
Title: An Open-Label, Dose-escalation, Phase I/IIa Study to Determine the Maximum Tolerated Dose, Recommended Dose, Efficacy, Pharmacokinetics and Pharmacodynamics of the Dual VEGFR-FGFR Tyrosine Kinase Inhibitor, E-3810, Given Orally as Single Agent to Patients With Advanced Solid Tumours
Brief Title: Study of Oral Lucitanib (E-3810), a Dual VEGFR-FGFR Tyrosine Kinase Inhibitor, in Patients With Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institut de Recherches Internationales Servier (Other)
Responsible Party: Sponsor
Organization: Servier (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E-3810-I-01
Record Dates: First submitted 2011-01-25; First posted 2011-01-26 (Estimated); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Solid Tumors
Keywords: VEGFRs; FGFR1; angiogenesis
MeSH Terms: interventions — E-3810

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lucitanib (Experimental)
  Interventions: Drug: Lucitanib

INTERVENTIONS:
Drug: Lucitanib — Oral administration, once daily (qd), in fasting conditions.
  Dose escalation - continuous schedule
  Dose expansion - continuous or intermittent dosing schedules (i.e. 5 days on/2days off or 21 days on/7 days off)
  Dosage form: hard gelatin capsules for oral administration (2.5, 5, 10, 30 and 50 mg strengths)
  Other Names: E-3810

SUMMARY:
Co-selective inhibition of VEGFRs and FGFR has the potential benefit of blocking the two most relevant players in tumor angiogenesis and simultaneously targeting proliferation in FGF-driven tumors. Lucitanib is a novel dual-targeted small molecule inhibitor of VEGFR1, 2, 3 and FGFR1 showing strong anti-angiogenic and anti-tumor activity in preclinical models at well-tolerated oral doses, with a favorable pharmacokinetic profile. These properties make it an attractive candidate for development in humans.

This is an open-label, uncontrolled, non-randomized, PhaseI/IIa study and its primary objective is to determine the Maximum Tolerated Dose (MTD) of Lucitanib administered orally, once daily, on a continuous schedule over the initial 28-day cycle.

Secondary objectives are to determine the safety profile, pharmacokinetics, pharmacodynamics and antitumour activity of Lucitanib, given as a single agent to adult patients with advanced solid tumours.

The study consists of two phases, a dose escalation phase followed by a dose-expansion phase at the identified Recommended Dose (RD). Eligible patients have histologically or cytologically confirmed locally advanced or metastatic solid tumours, relapsed or refractory to standard therapy. For the dose expansion, patients should have tumours bearing FGFR1 or 11q 12-14 amplification, assessed by FISH or CGH array, or "sensitive" to antiangiogenic treatment. These latter are defined as patients who have relapsed after having experienced stable disease (lasting at least six months) or partial response with prior treatment with an approved antiangiogenic regimen or patients with tumour types known to be potentially responsive to antiangiogenic agents but without such pretreatment if no antiangiogenic agents were approved and/or available for that specific condition (e.g thyroid cancer, thymic carcinoma).

Serial safety assessments, including evaluation of symptoms, physical examination and blood and urine laboratory analyses are performed throughout the study. Cardiac functions and blood pressure are monitored in consultation with a cardiologist. PK parameters are determined on plasma samples collected during the first 4-week cycle and analyzed using a validated LC-MS/MS method. Correlative studies include: (i) quantitative assessment of the effects of E-3810 on tumor vasculature by DCE-MRI and DCE-US imaging; (ii) assay of angiogenesis biomarkers i.e. soluble VEGFR2, VEGFR1, VEGF, bFGF, Collagen IV, FGF23 and PIGF(by ELISA) and circulating endothelial and progenitors cells (CEC and CEP). Tumor response is based on imaging according to RECIST; circulating tumor cells (CTC) are measured by the immunomagnetic CellSearch method.

In patients with tumours bearing FGFR1 amplifications the efficacy of Lucitanib will be formally tested according to a phase IIa design (one-stage Flaming design, H0=0.05, H1=0,30, power 0,80.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Histologically or cytologically confirmed, locally advanced or metastatic solid tumour, relapsed or refractory to standard therapy.

   In addition, only for the dose-expansion phase:

   i) solid tumour bearingFGFR1 amplification and, if breast cancer, with at least one prior endocrine therapy in the metastatic setting if ER+, and at least one chemotherapy line otherwise or ii) solid tumour progressing after having experienced SD (lasting for at least six month) or PR as best response to prior treatment with an approved or investigational antiangiogenic drug (e.g.: sorafenib, sunitinib, bevacizumab) as a single agent or in a chemotherapy combination or iii) solid tumour potentially sensitive to antiangiogenic treatments provided no antiangiogenic agents are approved and\or available for that specific condition.
3. Life expectancy ≥ 3 months
4. Full recovery (to Grade ≤ 1) from any prior surgical procedure(s) and from reversible side effects of prior therapy for cancer including radiation therapy, chemotherapy, and immunotherapy
5. Adequate haematologic function (haemoglobin ≥ 9 g/dL, absolute neutrophil count [ANC] ≥ 1500/mL, platelets ≥ 100,000/mL), adequate renal function (serum creatinine< 1.5 mg/dL or creatinine clearance > 40 mL/min), and adequate hepatic function (serum bilirubin ≤ 1.5 x upper limit of normal (ULN) mg/dL, aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≤ 3 x ULN)
6. Eastern Co-operative Oncology Group (ECOG) performance status ≤ 1
7. Negative serum pregnancy test at screening in women of childbearing potential
8. For men and women of child-bearing potential, use of a medically accepted method of contraception (abstinence, barrier method with spermicide, intrauterine device, or steroidal contraceptive for women and barrier method for men) for the duration of the study and for 60 days after participation in the study
9. Willingness and ability to give written informed consent and to comply with study procedures

Exclusion Criteria:

1. Active central nervous system (CNS) metastases not controlled by prior surgery or radiotherapy and/or low dose steroids
2. Haematologic malignancies (including leukaemia of any form, lymphoma, and multiple myeloma)
3. Active second malignancy or history of another malignancy within 2 years, with the exception of non-melanoma skin cancers or carcinoma in situ (CIS) of the breast or cervix or controlled, superficial carcinoma of the bladder
4. Treatment with any anticancer agent within 3 weeks, including investigational agents, chemotherapy, immunotherapy, biologic or hormonal therapy, surgery or radiation therapy (6 weeks for nitrosoureas, mitomycin or bevacizumab); luteinizing hormone releasing hormone (LHRH) agonist for prostate and mitotane for adrenal carcinoma are allowed.
5. Significant cardiovascular disease or condition, including:

   * Congestive heart failure requiring therapy
   * Ventricular and/or supra-ventricular arrhythmia requiring therapy
   * Severe conduction disturbance (including QTc interval prolongation > 0.47 sec [corrected], history of severe arrhythmia, or history of familial arrhythmia [e.g., Wolff-Parkinson-White syndrome])
   * Angina pectoris requiring therapy
   * Left ventricular ejection fraction (LVEF) < 50% evaluated by cardiac ultrasound (ECHO) or Multi Gated Acquisition Scan (MUGA)
   * Uncontrolled hypertension (defined as systolic blood pressure ≥ 140 mm Hg and/or diastolic blood pressure ≥ 90 mm Hg with optimized antihypertensive therapy)
   * Myocardial infarction (MI) within 6 months prior to administration of the first dose
   * > Class I cardiovascular disease according to the New York Heart Association's (NYHA) Functional Criteria
6. Ongoing treatment with Warfarin
7. Unavoidable concomitant treatment with any drug known for potential risk of causing Torsades de Pointes (see list in Appendix 4)
8. Significant gastrointestinal abnormalities, including ulcerative colitis, chronic diarrhoea associated with intestinal malabsorption, Crohn's disease, and/or prior surgical procedures affecting absorption or requirement for intravenous (IV) alimentation
9. Known pre-existing clinically significant disorder of the hypothalamic-pituitary axis, thyroid and adrenal gland
10. Serious/active bacterial, viral or fungal infection (including known active human immunodeficiency virus [HIV] infection) requiring systemic treatment
11. Concurrent severe or uncontrolled medical disease or organ system dysfunction which, in the opinion of the Investigators, would limit life expectancy to < 3 months, compromise the patient's safety, or interfere with evaluation of the safety of the investigational product
12. Psychiatric disorder or altered mental status that would preclude understanding of the informed consent process and/or completion of the necessary study procedures
13. Known hypersensitivity to gelatin or lactose monohydrate
14. Difficulty with swallowing
15. Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2010-07; Primary Completion 2016-09 (Actual); Study Completion 2017-05-04 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | First 4-week treatment cycle
Objective response rate (CR and PR according to RECIST) and rate of non-progressive disease at 24 weeks | Throughout the treatment period (tumor evaluation every 8 weeks)
  To be assessed only in patients with tumours bearing FGFR1 amplification.

SECONDARY OUTCOMES:
Pharmacokinetics following single and multiple dose administration | first 4-week treatment cycle
Tumor perfusion measured by DCE MRI and DCE-US | First 4-week treatment cycle
Circulating markers of angiogenesis: VEGFR2, VEGFR1, VEGF, Collagen IV, bFGF, CEC and CEP | First 4-week treatment cycle
Tumor response according to RECIST; CTC | Throughout the treatment period
Safety profile and dose limiting toxicities (DLT) | Troughout the treatment period
Free tumor circulating DNA | First 4-week treatment cycle

CONTACTS AND LOCATIONS:
Locations (4):
- France (2):
  - Institute Gustave Roussy, Villejuif, Paris
  - Hopital Louis Pradel, Lyon
- European Institute of Oncology, Milan, Italy
- Vall d' Hebron University Hospital, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Researchers can ask for a study protocol, patient-level and/or study-level clinical trial data including clinical study reports (CSRs).
  They can ask all interventional clinical studies:
  * submitted for new medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * Where Servier or an affiliate are the Marketing Authorization Holders (MAH). The date of the first Marketing Authorization of the new medicine (or the new indication) in one of the EEA Member States will be considered within this scope.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorisation in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.
URL: http://clinicaltrials.servier.com

REFERENCES:
- [Background] Liao M, Zhou J, Wride K, Lepley D, Cameron T, Sale M, Xiao J. Population Pharmacokinetic Modeling of Lucitanib in Patients with Advanced Cancer. Eur J Drug Metab Pharmacokinet. 2022 Sep;47(5):711-723. doi: 10.1007/s13318-022-00773-w. Epub 2022 Jul 18. PMID 35844029
- [Result] Soria JC, DeBraud F, Bahleda R, Adamo B, Andre F, Dientsmann R, Delmonte A, Cereda R, Isaacson J, Litten J, Allen A, Dubois F, Saba C, Robert R, D'Incalci M, Zucchetti M, Camboni MG, Tabernero J. Phase I/IIa study evaluating the safety, efficacy, pharmacokinetics, and pharmacodynamics of lucitanib in advanced solid tumors. Ann Oncol. 2014 Nov;25(11):2244-2251. doi: 10.1093/annonc/mdu390. Epub 2014 Sep 5. PMID 25193991